CLINICAL TRIAL: NCT03880084
Title: Longitudinal Assessment of Delirium, Agitation/Sedation, Pain and Dyspnea in Patients Admitted to Respiratory Intensive Care Unit for Acute Respiratory Failure (NIVILIUM)
Brief Title: Delirium, Agitation/Sedation, Pain and Dyspnea in Respiratory Intensive Care Unit (NIVILIUM)
Acronym: NIVILIUM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Alessandro Marchioni, Principal Investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio 5
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Failure; Delirium; Agitation,Psychomotor; Pain; Dyspnea; Mechanical Ventilation Complication
MeSH Terms: conditions — Respiratory Insufficiency; Delirium; Psychomotor Agitation; Pain; Dyspnea | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — To systematically assess the onset of delirium, quantify the level of agitation/sedation, estimate the grade of pain and survey the level of dyspnea in patients undergoing non invasive mechanical ventilation

SUMMARY:
Non-Invasive Mechanical Ventilation (NIV) has been increasingly used in the treatment of acute respiratory failure. Notwithstanding failure rates still remains high, ranging from 5% to 60%. The onset of delirium, agitation, pain and dyspnea may contribute to reduce the success rate of non invasive ventilation treatment. The aim of this study is to assess the incidence and impact of delirium, agitation, pain and dyspnea on clinical outcomes in a population of patient admitted to Respiratory Intensive Care Unit undergoing Non-Invasive Mechanical Ventilation for Acute Respiratory Failure.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute respiratory failure admitted to the Respiratory Intensive Care Unit of the University Hospital of Modena undergoing non invasive mechanical ventilation

Exclusion Criteria:

* age lower than 18
* Glasgow Coma Scale lower than 10 within 24 hours from Respiratory Intensive Care Unit admission
* need for immediate orotracheal intubation
* pregnancy
* previously established psychiatric disease or dementia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory failure admitted to the Respiratory Intensive Care Unit of the University Hospital of Modena undergoing non invasive mechanical ventilation not known for psychiatric disease or dementia
Sampling Method: Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium | 7 days from Respiratory Intensive Care Unit admission
  The onset of delirium will be assessed through the Confusion Assessment Method for Intensive Care Unit 7 scale, ranges 0-7, values > 2 indicate the presence of delirium
Incidence of agitation | 7 days from Respiratory Intensive Care Unit admission
  The onset of delirium will be assessed through the Richmond Agitation Sedation Scale ranges +4 to -5, values > 0 indicate the presence of agitation, values < 0 indicate the presence of sedation
Incidence of pain | 7 days from Respiratory Intensive Care Unit admission
  The onset of delirium will be assessed through the Behavioral Pain Scale, ranges 3-12, values > 4 indicate the presence of pain
Incidence of dyspnea | 7 days from Respiratory Intensive Care Unit admission
  The onset of delirium will be assessed through the Borg scale, ranges 0-10, values > 0 indicate the presence of dyspnea

SECONDARY OUTCOMES:
The impact of delirium on Non Invasive Ventilation Success | 30 days from Respiratory Intensive Care Unit admission
  The correlation between the onset of delirium and the failure rates of Non Invasive Ventilation Treatment will be assessed
The impact of agitation on Non Invasive Ventilation Success | 30 days from Respiratory Intensive Care Unit admission
  The correlation between the onset of agitation and the failure rates of Non Invasive Ventilation Treatment will be assessed
The impact of pain on Non Invasive Ventilation Success | 30 days from Respiratory Intensive Care Unit admission
  The correlation between the onset and level of pain and the failure rates of Non Invasive Ventilation Treatment will be assessed
The impact of dyspnea on Non Invasive Ventilation Success | 30 days from Respiratory Intensive Care Unit admission
  The correlation between the onset and level of dyspnea and the failure rates of Non Invasive Ventilation Treatment will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided